CLINICAL TRIAL: NCT04936386
Title: Knowledge and Perspective of Healthcare Professionals Related to Female Genital Mutation: a Regional Survey
Brief Title: Knowledge and Perspective of Healthcare Professionals About Female Genital Mutation
Acronym: FMG-HCPROF
Status: Completed | Type: Observational
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, Clinical Professor, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: FMG-HEALTHCAREPROF-SURVEY
Record Dates: First submitted 2021-06-19; First posted 2021-06-23 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Female Genital Mutilation Type I Status; Female Genital Mutilation Type II Status; Female Genital Mutilation Type III Status
Keywords: female genital mutilation; healthcare professionals
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals: Healthcare professionals (medical specialists and general practitioners, medical residents, midwives, professional nurses, medical students).
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — The survey is composed of 4 different sections: the first section included questions about demographic data of participants; the second part evaluated responders' knowledge about FGM; the third section focused on participants' working experience with patients affected by FGM and personal attitude related to this topic.

SUMMARY:
Each year over three million girls are at risk of being subjected to female genital mutilation (FGM) in several African countries. This regional survey aims to evaluate knowledge and perspective of healthcare professionals related to FGM.

DETAILED DESCRIPTION:
The survey iscomposed of 4 different sections: the first section included questions about demographic data of participants; the second part evaluated responders' knowledge about FGM; the third section focused on participants' working experience with patients affected by FGM and personal attitude related to this topic.

ELIGIBILITY:
Inclusion Criteria:

* medical specialists
* general medical practicians
* medical residents
* midwives
* professional nurses
* medical students
* residence in Liguria (Italy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthcare professionals working in Genoa
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Mean score related to knowledge about FGM | Baseline
  10-point score (0:minimal knowledge; 10: extensive knowledge) related to the knowledge of responders about FGM
Proportion of responders with active role in contrasting the procedures | Baseline
  Evalution of the personale attitude of responders to the topic (active role in contrasting the procedures)
Proportion of responders feeling confortable in treating patients affected | Baseline
  Evalution of the personale attitude of responders to the topic (responders feeling confortable in treating patients affected)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdulcadir J, Catania L, Hindin MJ, Say L, Petignat P, Abdulcadir O. Female Genital Mutilation: A Visual Reference and Learning Tool for Health Care Professionals. Obstet Gynecol. 2016 Nov;128(5):958-963. doi: 10.1097/AOG.0000000000001686. PMID 27741194